CLINICAL TRIAL: NCT02011633
Title: An Open-label, Randomized, Single-dose Crossover Study to Compare the Pharmacokinetics After the Administration of HCP1201 Tablet 500/10 mg and Coadministration of Metformin SR 500 mg and Rosuvastatin 10 mg in Healthy Volunteers
Brief Title: Comparison of PK After Administration of HCP1201 and Co-administration of Metformin SR 500mg and Rosuvastatin 10mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-MERO-105
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HCP1201, Part 1 (Experimental): Participants received a single oral dose of the HCP1201 500/10 mg under fasting condition, on Period 1(for participants randomized to Sequence 1) or on Period 2(for participants randomized to Sequence 2).
  Interventions: Drug: HCP1201 500/10mg
- Metformin and Rosuvastatin, Part1 (Active Comparator): Participants received a single oral dose of coadministration of Metformin SR 500 mg and Rosuvastatin 10 mg under fasting condition, on Period 1(for participants randomized to Sequence 1) or on Period 2(for participants randomized to Sequence 2).
  Interventions: Drug: Metformin SR 500mg; Drug: Rosuvastatin 10mg
- HCP1201, Part 2 (Experimental): Participants received a single oral dose of the HCP1201 500/10mg under fed condition, on Period 1(for participants randomized to Sequence 1) or on Period 2(for participants randomized to Sequence 2).
  Interventions: Drug: HCP1201 500/10mg
- Metformin and Rosuvastatin, Part 2 (Active Comparator): Participants received a single oral dose of coadministration of Metformin SR 500mg and Rosuvastatin 10mg under fed condition, on Period 1(for participants randomized to Sequence 1) or on Period 2(for participants randomized to Sequence 2).
  Interventions: Drug: Metformin SR 500mg

INTERVENTIONS:
Drug: HCP1201 500/10mg — 500mg Metformin/10mg rosuvastatin fixed dose combination tablet orally in the morning on day1 or day8.
  Arms: HCP1201, Part 1; HCP1201, Part 2
Drug: Metformin SR 500mg — Co-administration of Metformin 500mg and Rosuvastatin 10mg orally in the morning on day1 or day8.
  Other Names: Glucophage SR 500 mg
  Arms: Metformin and Rosuvastatin, Part 2; Metformin and Rosuvastatin, Part1
Drug: Rosuvastatin 10mg — Co-administration of Metformin 500mg and Rosuvastatin 10mg orally in the morning on day1 or day8.
  Other Names: Crestor 10mg
  Arms: Metformin and Rosuvastatin, Part1

SUMMARY:
To compare the pharmacokinetic characteristics between HCP1201 tablet 500/10 mg and co-administration of metformin 500 mg plus rosuvastatin 10 mg under fasted and fed state, respectively.

DETAILED DESCRIPTION:
An Open-label, Randomized, Single-dose Crossover Study to Compare the Pharmacokinetics After the Administration of HCP1201 Tablet 500/10 mg and Coadministration of Metformin SR 500 mg and Rosuvastatin 10 mg in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer, age 20~55 years
* The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 27 kg/m2
* Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial.

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study
* History of relevant drug allergies or clinically significant hypersensitivity reaction.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
metformin, rosuvastatin Cmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
metformin, rosuvastatin AUClast | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h

SECONDARY OUTCOMES:
Metformin, rosuvastatin Tmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin T1/2 | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin AUCinf | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Wooseong Huh, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea